CLINICAL TRIAL: NCT02224144
Title: A Comparative Trial of Calcitriol Versus Placebo for the Preservation of Bone Mass and Strength After Kidney Transplantation
Brief Title: Bone Mass and Strength After Kidney Transplantation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: Satellite Healthcare (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: AAAM7850
Record Dates: First submitted 2014-08-22; First posted 2014-08-25 (Estimated); Results first posted 2025-03-07 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: End Stage Renal Disease; Kidney Transplantation; Bone Loss; Fractures; Vascular Calcifications
Keywords: Kidney Transplantation; Calcitriol; Bone Mineral Density; Bone Mass and Strength; Vascular Calcifications; Hyperparathyroidism; Parathyroid Hormone
MeSH Terms: conditions — Kidney Failure, Chronic; Bone Diseases, Metabolic; Fractures, Bone; Vascular Calcification; Hyperparathyroidism | interventions — Cholecalciferol; Calcitriol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Vitamin D3 plus Calcitriol (Experimental): 1 pill of Vitamin D3 (cholecalciferol) 1000 IU daily for 12 months
  1 pill of Rocaltrol (calcitriol) 0.5 mcg daily for 12 months
  Interventions: Drug: Vitamin D3; Drug: Calcitriol
- Vitamin D3 plus Placebo (Placebo Comparator): 1 pill of Vitamin D3 (cholecalciferol) 1000 IU per day for 12 months
  1 pill of placebo (sugar pill) per day for 12 months
  Interventions: Drug: Vitamin D3; Drug: Placebo

INTERVENTIONS:
Drug: Vitamin D3 — Vitamin D3 1000 IU per day for 12 months
  Other Names: cholecalciferol
Drug: Calcitriol — Calcitriol (Rocaltrol) 0.5 mcg per day for 12 months
  Other Names: Rocaltrol
  Arms: Vitamin D3 plus Calcitriol
Drug: Placebo — Placebo (sugar pill) 1 pill per day for 12 months
  Arms: Vitamin D3 plus Placebo

SUMMARY:
The purpose of this study is to test whether active vitamin D (calcitriol) protects bones from weakening and protects blood vessels from calcium deposits over the first year of kidney transplantation.

DETAILED DESCRIPTION:
Kidney transplant recipients at highest fracture risk, as determined by epidemiologic studies (Caucasians and older recipients). Rocaltrol (calcitriol) is a synthetic vitamin D analog which is active in the regulation of the absorption of calcium from the gastrointestinal tract and its utilization in the body.

ELIGIBILITY:
Inclusion Criteria:

* Age older than 18
* Self-describes as White race

Exclusion Criteria:

* Lower extremity amputations
* Non-ambulatory
* Paget´s disease of bone
* Current hyperthyroidism, untreated hypothyroidism
* Medical diseases (end stage liver, intestinal malabsorption)
* Use within the prior year pod anti-seizure medications that induce the cytochrome P450 system, testosterone, estrogen, selective estrogen receptor modulators
* Weight >300 pounds
* Dual organ transplant
* Myocardial infarction or stroke
* Tobacco use within the past year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2014-08-18 (Actual); Primary Completion 2016-10-12 (Actual); Study Completion 2016-10-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Nickolas, MD, MS, Principal Investigator — Columbia University
Locations (1):
- Columbia University Irving Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Iyer SP, Nikkel LE, Nishiyama KK, Dworakowski E, Cremers S, Zhang C, McMahon DJ, Boutroy S, Liu XS, Ratner LE, Cohen DJ, Guo XE, Shane E, Nickolas TL. Kidney transplantation with early corticosteroid withdrawal: paradoxical effects at the central and peripheral skeleton. J Am Soc Nephrol. 2014 Jun;25(6):1331-41. doi: 10.1681/ASN.2013080851. Epub 2014 Feb 7. PMID 24511131

RESULTS

PARTICIPANT FLOW:
Groups:
- Vitamin D3 Plus Calcitriol: Participants will take 1000 IU of Vitamin D3 (cholecalciferol) and 0.5 mcg of Rocaltrol (calcitriol) daily for 12 months.
- Vitamin D3 Plus Placebo: Participants will take 1000 IU of Vitamin D3 (cholecalciferol) and 1 sugar pill (placebo) daily for 12 months.
Period: Overall Study
Arm/Group | Vitamin D3 Plus Calcitriol | Vitamin D3 Plus Placebo
Started | 32 | 29
Completed | 27 | 27
Not Completed | 5 | 2
Not completed — Lost to Follow-up | 3 | 1
Not completed — Death | 2 | 0
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vitamin D3 Plus Calcitriol | Vitamin D3 Plus Placebo | Total
Number analyzed (Participants) | 32 | 29 | 61
Age, Continuous [Mean (Standard Deviation); unit: years] | 51 (14) | 51 (13) | 51 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 9 | 20
  Male | 21 | 20 | 41
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 32 | 28 | 60
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 32 | 29 | 61

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Bone Density From Pre to Post-calcitriol Treatment Compared to Placebo as Assessed by Both Standard Methodologies
Description: Novel high resolution bone imaging can separately measure and quantify cortical and trabecular responses to bone active treatments. Finite element analysis (FEA) can be applied to HRpQCT datasets. to provide a computational estimate of bone mechanical competence that has been validated against true compressive tests of bone stiffness and strength.
Time Frame: Baseline, 12 months
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Vitamin D3 Plus Calcitriol | Vitamin D3 Plus Placebo
Number analyzed (Participants) | 27 | 27
percent change | -0.81 (0.54) | -0.70 (0.46)

2. Secondary Outcome: Percent Change in Areal Bone Mass Density From Baseline to 12 Months After Transplantation
Description: Apply imaging methods to shed light on whether preservation of areal bone mineral density (BMD) measured by dual-energy x-ray absorptiometry (DXA) is accompanied by preservation of bone mechanical competence measured by a method that has been validated against true compressive tests of bone strength.
Time Frame: Baseline, 12 months
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Vitamin D3 Plus Calcitriol | Vitamin D3 Plus Placebo
Number analyzed (Participants) | 27 | 27
percent change
  BMD Lumbar Spine | 1.91 (0.94) | 0.85 (1.05)
  BMD Total Hip | 0.88 (0.94) | -0.09 (1.03)
  BMD Femoral Neck | 0.64 (1.31) | -0.45 (1.41)
  BMD Ultradistal Radius | -3.19 (1.15) | -3.30 (0.99)

3. Secondary Outcome: Percent Change in Failure Load Pre- and Post-transplantation Measured by High Resolution Imaging Methods
Description: Failure load refers to the maximum amount of force a bone can withstand before it fractures. Volumetric BMD and microarchitecture of cortical and trabecular compartments were measured using HR-pQCT first- (XCT1) and second-generation scanners (XCT2), with voxel size 82 μm and 60 μm respectively. HR-pQCT imaging was performed on the non-dominant radius and tibia.
Time Frame: Baseline, 12 months
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Vitamin D3 Plus Calcitriol | Vitamin D3 Plus Placebo
Number analyzed (Participants) | 27 | 27
percent change
  Scan of radius | -5 (1) | -3.4 (1.3)
  Scan of tibia | -1.9 (1.2) | -2.5 (1.9)

4. Secondary Outcome: Percent Change of Cortical Porosity Pre- and Post-intervention
Description: Cortical porosity was calculated as the percentage of void space in the cortex. HR-pQCT imaging was performed on the non-dominant radius and tibia.
Time Frame: Baseline, 12 months
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Vitamin D3 Plus Calcitriol | Vitamin D3 Plus Placebo
Number analyzed (Participants) | 27 | 27
percent change
  Scan of radius | 11.6 (11.1) | 12.5 (7.8)
  Scan of tibia | 21 (7) | 13.3 (5.6)

5. Secondary Outcome: Percent Change in Vascular Calcifications Loads of the Lower Extremity
Description: A semi-automated algorithm implemented in image processing language was used for assessment of lower leg arterial calcification (LLAC) and wrist arterial calcification (WAC).
Time Frame: Baseline, 12 months
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Vitamin D3 Plus Calcitriol | Vitamin D3 Plus Placebo
Number analyzed (Participants) | 27 | 27
percent change
  LLAC | 1.5 (3.5) | -8.4 (6.1)
  WAC | 112 (118) | 68 (70)

6. Secondary Outcome: Number of Patients With Vascular Calcifications of the Lower Extremity
Description: Quantification of calcifications of the anterior and posterior tibia arteries measured by a novel method applied to HRpQCT at baseline and 12 months.
Time Frame: Baseline, 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Vitamin D3 Plus Calcitriol | Vitamin D3 Plus Placebo
Number analyzed (Participants) | 27 | 27
Participants
  Baseline | 13 | 9
  12 months | 13 | 8

7. Secondary Outcome: Percent Change in Pre- and Post- Intervention Parathyroid Hormone (PTH) Levels
Description: PTH levels were measured in participants to confirm the hypothesis that calcitriol administration over the first year of kidney transplantation would protect the cortical skeleton in recipients managed without corticosteroids due to its ability to suppress PTH and bone remodeling.
Time Frame: Baseline, 12 months
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Vitamin D3 Plus Calcitriol | Vitamin D3 Plus Placebo
Number analyzed (Participants) | 27 | 27
percent change | -63 (11) | -59 (6)

8. Secondary Outcome: Percent Change in Pre- and Post- Intervention Levels of Bone Remodeling Markers for Bone Remodeling Assessment
Description: Participants underwent a blood draw for measurement of bone markers: bone-specific alkaline phosphatase (BSAP), propeptide of type 1 procollagen (P1NP), osteocalcin (OC), and the bone resorption marker serum cross-linked C-telopeptide of type I collagen (CTX).
Time Frame: Baseline, 12 months
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Vitamin D3 Plus Calcitriol | Vitamin D3 Plus Placebo
Number analyzed (Participants) | 27 | 27
percent change
  BSAP | 9.6 (13.2) | 60 (35)
  Osteocalcin | -80 (4) | -72 (6.2)
  P1NP | -14 (23) | 2.9 (17.7)
  CTX | -77 (5) | -70 (6)

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Vitamin D3 Plus Calcitriol | Vitamin D3 Plus Placebo
All-Cause Mortality (participants affected / at risk) | 2/32 | 0/29
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/29
Other Adverse Events (participants affected / at risk) | 12/32 | 8/29
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Vitamin D3 Plus Calcitriol (N=32) | Vitamin D3 Plus Placebo (N=29)
Hypercalcemia (Musculoskeletal and connective tissue disorders) | 12 | 1
Rejection (Surgical and medical procedures) | 4 | 8
Fracture after transplantation (Musculoskeletal and connective tissue disorders) | 0 | 2
Hospitalizations (General disorders) | 9 | 7
Calcifications on Kidney Biopsy (Renal and urinary disorders) | 7 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes